CLINICAL TRIAL: NCT01448278
Title: Pain Evaluation After ACL Ligamentoplasty: "All-inside" Versus Classical Technique. A Prospective Randomised Comparative Study
Brief Title: Pain Evaluation After Anterior Cruciate Ligament (ACL) Ligamentoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Shahnaz Klouche, MD, Physician Responsible of Clinical Research, Hospital Ambroise Paré Paris
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: APR112010
Record Dates: First submitted 2011-10-04; First posted 2011-10-07 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Arthroscopic Anterior Cruciate Ligament Reconstruction
Keywords: Anterior cruciate ligament; Arthroscopy; Incomplete bone tunnels; Anterior cruciate ligament reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- All-inside technique (Experimental)
  Interventions: Procedure: "All-inside"
- Classical technique (Active Comparator)
  Interventions: Procedure: Classical technique

INTERVENTIONS:
Procedure: "All-inside" — The "All-inside" technique is a new minimally invasive procedure for anterior cruciate ligament reconstruction (ACL). It consists of incomplete bone tunnels drilling and cortical fixation.
  Arms: All-inside technique
Procedure: Classical technique — The Classical technique is a usual procedure for anterior cruciate ligament reconstruction (ACL). The fixation is achieved with interference screws.
  Arms: Classical technique

SUMMARY:
The "All-inside" method is a new minimally invasive procedure for anterior cruciate ligament reconstruction (ACL). It consists of incomplete bone tunnels drilling and cortical fixation. In the so-called "classical" method, the fixation is achieved with interference screws.

The hypothesis of this study was that the "All-inside" technique causes less pain than the conventional technique. The main objective was to evaluate the immediate postoperative pain for the first ten days and at one month from the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Total or partial tear of the Anterior Cruciate Ligament

Exclusion Criteria:

* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Pain assessment on a Visual Analogical Scale | One month after surgery

SECONDARY OUTCOMES:
Pain assessment on a Visual Analogical Scale | First ten days
Analgesics consumption | First ten days
Functional evaluation with IKDC score | Change from base-line in IKDC objective score at 6 months
Discharge of crutches and orthesis | Time frame from surgery
Radiographic analysis of tunnels positioning according to Aglietti's criteria | One month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Hardy, Ph.D., Principal Investigator — Hospital Ambroise Paré Paris; Horea Benea, MD, Study Director — Ambroise Paré Hospital; Henri d'Astorg, MD, Study Director — Ambroise Paré Hospital
Locations (1):
- Ambroise Paré Hospital, Boulogne-Billancourt, Île-de-France Region, France

REFERENCES:
- [Derived] Benea H, d'Astorg H, Klouche S, Bauer T, Tomoaia G, Hardy P. Pain evaluation after all-inside anterior cruciate ligament reconstruction and short term functional results of a prospective randomized study. Knee. 2014 Jan;21(1):102-6. doi: 10.1016/j.knee.2013.09.006. Epub 2013 Oct 5. PMID 24269603